CLINICAL TRIAL: NCT03237390
Title: Phase I Study of CDK4/6 Inhibitor Ribociclib (LEE011) Combined With Gemcitabine in Patients With Advanced Solid Tumors
Brief Title: Ribociclib and Gemcitabine Hydrochloride in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1613; NCI-2017-01316 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1613 (Other: Mayo Clinic)
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Gemcitabine; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gemcitabine hydrochloride, ribociclib) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and ribociclib PO QD on days 8-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ribociclib

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011

SUMMARY:
This phase I trial studies the side effects and best dose of ribociclib and gemcitabine hydrochloride in treating patients with solid tumors that have spread to other places in the body. Ribociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ribociclib and gemcitabine hydrochloride may work better in treating patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the dose-limiting toxicities and identify the maximum tolerated dose (MTD) and recommended phase II dose of the combination of ribociclib and gemcitabine hydrochloride (gemcitabine) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To describe the safety and tolerability of the combination of ribociclib and gemcitabine.

II. To describe the pharmacokinetic (PK) of ribociclib in combination with gemcitabine.

III. To describe preliminary evidence of efficacy of the combination of ribociclib and gemcitabine.

TERTIARY OBJECTIVES:

I. To evaluate the correlation of CDK4/6, cyclin D1 and cyclin D3 amplification, retinoblastoma (RB) and P16 expression in archived and biopsied tumor tissue with treatment response.

OUTLINE: This is a dose-escalation study.

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8 and ribociclib orally (PO) once daily (QD) on days 8-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/metastatic solid malignancy for which no standard treatment option exists that will confer clinical benefit
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Dose expansion phase only: must have at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Ability to provide written informed consent which must be obtained prior to any screening procedures and according to local guidelines
* Life expectancy of >= 12 weeks
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Potassium >= lower limit of normal (LLN) range for the institution
* Calcium >= LLN (corrected for serum albumin, if albumin abnormal)
* Magnesium >= LLN
* Sodium >= LLN
* Phosphorus >= LLN; NOTE: Supplementation may be given before the first dose of study medication
* International normalized ratio (INR) =< 1.5
* Serum creatinine =< 1.5 mg/dL or creatinine clearance >= 50 mL/min (calculated by Cockcroft Gault equation)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) or =< 5 x ULN if liver metastases are present
* Total bilirubin =< 3.0 x ULN; if patient has known Gilbert?s syndrome direct bilirubin =< 1.5 x ULN
* Standard 12-lead electrocardiography (ECG) with the following parameters at screening (defined as the mean of the triplicate ECGs):

  * Fridericia's correction formula (QTcF) interval at screening < 450 msec (using Fridericia? s correction)
  * Resting heart rate 50 to 100 beats per minute
* Negative pregnancy test performed =< 7 days prior to registration (women of childbearing potential only)
* Able to swallow ribociclib capsules
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide mandatory blood samples for research purposes

Exclusion Criteria:

* Previous anti-cancer chemotherapy, immunotherapy or investigational agents =< 28 days prior to registration
* Received radiotherapy =< 28 days or limited field radiation for palliation =< 14 days prior to registration, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom >= 25% of the bone marrow was irradiated
* Major surgery =< 14 days prior to registration or has not recovered from major side effects (tumor biopsy is not considered as major surgery)
* Active clinically serious infections or other serious uncontrolled medical conditions
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Baseline neuropathy of > grade 2
* Known hypersensitivity to any of the excipients of ribociclib
* Known human immunodeficiency virus (HIV) patients with active and untreated disease
* Central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * >= 28 days from prior therapy completion (including radiation and/or surgery) to registration
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
* Clinically significant, uncontrolled heart disease and/ or cardiac repolarization abnormalities including any of the following:

  * History of unstable angina pectoris, symptomatic pericarditis, myocardial infarction, coronary artery bypass grafting or coronary angioplasty =< 12 months prior to registration
  * History of documented congestive heart failure (New York Heart Association functional classification III - IV)
  * Documented cardiomyopathy
  * Left ventricular ejection fraction (LVEF) < 50% as determined by echocardiogram (ECHO)
  * Clinically significant cardiac arrhythmias ( e.g ventricular tachycardia) , left bundle branch block, high-grade atrioventricular (AV) block ( e.g bifascucular block, Mobitz type II and third degree AV block)
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for torsades de pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause torsades de pointe that cannot be discontinued (within 5 half-lives or =< 7 days prior to registration) or replaced by safe alternative medication
    * Inability to determine the QT interval on screening (QTcF, using Fridericia? s correction)
* Systolic blood pressure > 160 mmHg or < 90 mmHg
* Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator?s judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g., chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections etc.)
* Currently receiving any of the following medications and cannot be discontinued 7 days prior to starting the study

  * Herbal supplements including grapefruit, grapefruit hybrids, pummelos, star-fruit, Seville oranges or products containing the juice of each; orange juice is allowed
  * Known strong inducers or inhibitors of CYP3A4/5 including grapefruit, grapefruit hybrids, pomelos, star-fruit, and Seville oranges
  * Medications known to have a narrow therapeutic window and are predominantly metabolized through CYP3A4
* Currently receiving or has received systemic corticosteroids (=< 14 days prior to registration, or who have not fully recovered from side effects of such treatment); NOTE: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* History of non-compliance to medical regimen or inability to grant consent
* Currently receiving warfarin or other warfarin-derived anticoagulant for treatment, prophylaxis or otherwise; Note: Therapy with heparin, direct oral anticoagulants, low molecular weight heparin (LMWH) or fondaparinux is allowed
* Participation in a prior investigational study =< 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
* Failure to recover from all adverse events/toxicities related to prior anticancer therapies to grade 1 per National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.03; NOTE: Exception: patients with any grade of alopecia are allowed to enter the study
* Child-Pugh score B or C (for cirrhosis patients only)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation; highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening), the vasectomized male partner should be the sole partner for that patient
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
  * Note: In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment; Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction
  * Note: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse while taking the drug and for 21 days after stopping treatment and should not father a child in this period; Note: A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Known standard therapy for the patient?s disease that is potentially curative or definitely capable of extending life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 21 days
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least 2 patients (out of 6).

SECONDARY OUTCOMES:
Best response defined as best objective status recorded from the start of the treatment until disease progression/recurrence | Up to 18 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group). The number of responses may indicate further evaluation for specific tumor types in a phase II setting.
Confirmed response defined to be a stringent complete response, complete response, very good partial response, or partial response | Up to 18 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group). The number of responses may indicate further evaluation for specific tumor types in a phase II setting.
Incidence of adverse events | Up to 30 days after last dose
  Number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized. Adverse events that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal Common Toxicity Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence
Pharmacokinetic (PK) of ribociclib | Pre-ribociclib dose, 0.5, 1, 2, 4, 6, and 8 hours post dose on days 8 and 14 course 1 and pre-gemcitabine hydrochloride dose on day 1 course 2
  A population PK model will be developed utilizing the PK time points collected, and then used to estimate individual area under the curves or clearance of ribociclib in combination with gemcitabine hydrochloride. The effect of the combination on PK of each drug will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics.

OTHER OUTCOMES:
CDK2/4/6, Cyclin D1 and Cyclin D3 amplification, retinoblastoma (RB) and P16 expression | Up to 18 months
  CDK2/4/6, Cyclin D1 and Cyclin D3 amplification, RB and P16 expression in archived and biopsied tumor tissue with be correlated with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Norman A, Seetharam M, Allred J, Kong J, Opyrchal M, Ma WW, Lou Y, Dy GK, Mahipal A, Weroha SJ, Wahner Hendrickson AE, Reid JM, Adjei AA. A phase I study of the CDK4/6 inhibitor ribociclib combined with gemcitabine in patients with advanced solid tumors. BJC Rep. 2025 Jan 14;3(1):1. doi: 10.1038/s44276-024-00107-0. PMID 39809926
- [Derived] Seetharam M, Norman A, Allred J, Kong J, Opyrchal M, Ma WW, Lou Y, Dy GK, Mahipal A, Weroha J, Wahner-Hendrickson A, Reid JM, Adjei AA. A Phase I Study of sequences of the CDK4/6 Inhibitor, Ribociclib Combined with Gemcitabine in Patients with Advanced Solid Tumors. Res Sq [Preprint]. 2024 Apr 25:rs.3.rs-4261257. doi: 10.21203/rs.3.rs-4261257/v1. PMID 38746220
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials